CLINICAL TRIAL: NCT06306209
Title: Inflammatory Control of Antidepressant Efficacy: a Pharmaco-epigenetic Approach
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Sara Poletti, Principal Investigator, IRCCS Ospedale San Raffaele
Other Study IDs: DeFLAME
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Mood Disorders; Major Depressive Disorder
MeSH Terms: conditions — Mood Disorders; Depressive Disorder, Major | interventions — Therapeutics; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MDD: 80 patients with a depressive episode in course of major depression (MDD) and treated with SSRI's will be studied. The study does not include the evaluation of pharmacological treatments. The treatments will be administered in the judgment of the attending physician, independently of the experimental protocol.
  Interventions: Other: Treatment as usual (TAU), i.e., pharmacotherapy plus clinical management

INTERVENTIONS:
Other: Treatment as usual (TAU), i.e., pharmacotherapy plus clinical management — All participants enrolled in the study will receive Treatment as usual (TAU), i.e., pharmacotherapy plus clinical management. Clinicians will be free to choose antidepressant medication, doses and drug combinations, including augmentations strategies and non-pharmacological treatments, which will follow standard clinical treatment guidelines for MDD.

SUMMARY:
Major depressive disorder (MDD) is a chronic, recurring and potentially life-threatening illness that affects up to 10% of the population across the globe.It posits that the increase in serotonin levels induced by Selective Serotonin Reuptake Inhibitors (SSRIs) does not affect mood per se, but enhances brain plasticity and thus amplifies the influence of the environment on the individual. Thus, SSRI treatment has not a univocal effect but, in a favorable environment, it would lead to a reduction of symptoms while in a stressful environment might lead to a worse prognosis.Such innovative view opens new perspectives on how to improve SSRI efficacy by controlling the environment. However, often it is not possible to act on the quality of the living environment because of constraints due to patient's personal history and unchangeable life circumstances. In these cases, the pharmacological modulation of the factors underlying the link between living environment and SSRI efficacy represents a novel and desirable strategy to improve treatment outcome even in patients living in adverse conditions, which are very common in depressed patients. Inflammatory levels are markedly affected by the socioeconomic status and thus by the quality of the living environment. The hypothesis of the present project is that inflammation mediates the influence of the environment on SSRI outcome.Therefore, the control of inflammatory levels is a promising strategy to improve treatment efficacy and overcome the limited SSRI efficacy, especially when administered in patients living in adverse conditions. A further hypothesis is that the influence of the environment on inflammation, in turn affecting SSRI efficacy, occurs through epigenetic modifications. Therefore, the project aims at developing a pharmaco-epigenetic approach as effective treatment for MDD. In addition, through neuroimaging investigations, it will provide important information about functional and structural brain modifications associated to SSRI efficacy in patients.

Both males and females will be considered because MDD is twice as common in women than men, suggesting that different mechanisms may underlie the psychopathology in the two sexes.

ELIGIBILITY:
Inclusion Criteria:

A depressive episode according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria in the course of MDD with:

HDRS score > 17 Age 18-65 years; In treatment with SSRIs Signed informed consent, able to understand, speak and write the national language

Exclusion Criteria:

* History of bipolar disorder, schizophrenia, schizoaffective disorder, psychosis not otherwise specified; anorexia or bulimia nervosa;
* Taking following medications: antipsychotics, anticonvulsants, mood stabilizers; stimulants
* Active infection requiring antibiotics therapy;
* Immunosuppressed patient
* Other chronic diseases
* Signs of active infection requiring treatment
* Use of anti-inflammatory medication on a regular basis for a chronic inflammatory/autoimmune Disorder.
* Forbidden treatment: corticosteroids, Non Steroidal Anti-inflammatory Drugs, immunosuppressant IV-Ig based treatment
* Ongoing fever, infection treated by antibiotics or uncontrolled diabetes type I or II;
* Existing cancer or history of cancer in the last 5 years (except skin epidermoid cancer or in-situ cervix cancer);
* Known HIV infection or clinically manifest Acquired Immune Deficiency Syndrome (AIDS),
* Parkinson's or Alzheimer's disease, or any other serious condition likely to interfere e with the conduct of the trial;
* Abuse of drugs or alcohol in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are always informed on currently ongoing and upcoming (clinical) duties during their regular outpatient clinic visits and at the first interview during hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
The potential role of inflammation as the causal link between the quality of the environment and SSRI efficacy | Blood samples will be collected at baseline time and after 3 months in correspondence with routine blood sampling performed at the patients arrival in the hospital.
  we will measure the levels of peripheral inflammatory markers and implement mediation/moderation model to investigate if inflammatory markers mediate/moderate the association between the environment (number of stressful events) and SSRIs efficacy (response to treatment: 50% reduction at the hamilton depression rating scale (HDRS) - scores min 0 max 52, higher score higher severity).
interaction between early stress and recent stress on the response to treatment and the role of inflammation | at baseline, at 3 months follow up
  we will investigate whether patients exposed to early stress (Risk Families Questionnaire (RFQ) score min 13, max 65, higher scores higher exposure to early life events;Childhood Trauma Questionnaire (CTQ) score min 28, max 140, higher score higher childhood trauma) have higher levels of inflammatory markers and are more vulnerable to recent stress (number of events) and if this interaction affects the response to treatment (50% reduction at HDRS)
identification of neurobiological predictors of response to treatment | at baseline, at 3 months follow up
  MRI scans will be performed at baseline and 3 month followup (Functional MRI). Changes in gray matter volumes which predict response to treatment (50% reduction at HDRS)will be identified
identification of neurobiological predictors of response to treatment | at baseline, at 3 months follow up
  MRI scans will be performed at baseline and 3 month followup (Diffusion Tensor Imaging (DTI);) Changes in white matter microstructure (fractional anisotropy) which predict response to treatment (50% reduction at HDRS)will be identified
identification of neurobiological predictors of response to treatment | at baseline, at 3 months follow up, at 6 months follow up
  Changes in peripheral inflammatory markers and transcriptomic between baseline and follow-up able to predict response to treatment (50% reduction at HDRS) will be identified

SECONDARY OUTCOMES:
epigenetic changes in cytokine regulating genes which could mediate the effect of stress on response to treatment. | Blood samples will be collected at baseline time and after 3 months in correspondence with routine blood sampling performed at the patients arrival in the hospital.
  mediation/moderation models will be implemented to identify epigenetic changes (RNA sequencing) that mediate/moderate the association between recent stress (number of events) and response to treatment (50% reduction at HDRS)

CONTACTS AND LOCATIONS:
Overall Officials: sara Poletti, PhD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Background] Branchi I. The double edged sword of neural plasticity: increasing serotonin levels leads to both greater vulnerability to depression and improved capacity to recover. Psychoneuroendocrinology. 2011 Apr;36(3):339-51. doi: 10.1016/j.psyneuen.2010.08.011. Epub 2010 Sep 26. PMID 20875703
- [Background] Maya Vetencourt JF, Sale A, Viegi A, Baroncelli L, De Pasquale R, O'Leary OF, Castren E, Maffei L. The antidepressant fluoxetine restores plasticity in the adult visual cortex. Science. 2008 Apr 18;320(5874):385-8. doi: 10.1126/science.1150516. PMID 18420937
- [Background] Belsky J, Jonassaint C, Pluess M, Stanton M, Brummett B, Williams R. Vulnerability genes or plasticity genes? Mol Psychiatry. 2009 Aug;14(8):746-54. doi: 10.1038/mp.2009.44. Epub 2009 May 19. PMID 19455150
- [Background] Alboni S, van Dijk RM, Poggini S, Milior G, Perrotta M, Drenth T, Brunello N, Wolfer DP, Limatola C, Amrein I, Cirulli F, Maggi L, Branchi I. Fluoxetine effects on molecular, cellular and behavioral endophenotypes of depression are driven by the living environment. Mol Psychiatry. 2017 Apr;22(4):552-561. doi: 10.1038/mp.2015.142. Epub 2015 Sep 15. PMID 26645631
- [Background] Branchi I, Santarelli S, Capoccia S, Poggini S, D'Andrea I, Cirulli F, Alleva E. Antidepressant treatment outcome depends on the quality of the living environment: a pre-clinical investigation in mice. PLoS One. 2013 Apr 30;8(4):e62226. doi: 10.1371/journal.pone.0062226. Print 2013. PMID 23653679
- [Background] Chiarotti F, Viglione A, Giuliani A, Branchi I. Citalopram amplifies the influence of living conditions on mood in depressed patients enrolled in the STAR*D study. Transl Psychiatry. 2017 Mar 21;7(3):e1066. doi: 10.1038/tp.2017.35. PMID 28323288
- [Background] Cohen A, Houck PR, Szanto K, Dew MA, Gilman SE, Reynolds CF 3rd. Social inequalities in response to antidepressant treatment in older adults. Arch Gen Psychiatry. 2006 Jan;63(1):50-6. doi: 10.1001/archpsyc.63.1.50. PMID 16389196
- [Background] Iosifescu DV, Clementi-Craven N, Fraguas R, Papakostas GI, Petersen T, Alpert JE, Nierenberg AA, Fava M. Cardiovascular risk factors may moderate pharmacological treatment effects in major depressive disorder. Psychosom Med. 2005 Sep-Oct;67(5):703-6. doi: 10.1097/01.psy.0000170338.75346.d0. PMID 16204427
- [Background] Alley DE, Seeman TE, Ki Kim J, Karlamangla A, Hu P, Crimmins EM. Socioeconomic status and C-reactive protein levels in the US population: NHANES IV. Brain Behav Immun. 2006 Sep;20(5):498-504. doi: 10.1016/j.bbi.2005.10.003. Epub 2005 Dec 2. PMID 16330181
- [Background] Miller AH, Maletic V, Raison CL. Inflammation and its discontents: the role of cytokines in the pathophysiology of major depression. Biol Psychiatry. 2009 May 1;65(9):732-41. doi: 10.1016/j.biopsych.2008.11.029. Epub 2009 Jan 15. PMID 19150053
- [Background] Miller AH, Raison CL. The role of inflammation in depression: from evolutionary imperative to modern treatment target. Nat Rev Immunol. 2016 Jan;16(1):22-34. doi: 10.1038/nri.2015.5. PMID 26711676
- [Background] Raison CL, Rutherford RE, Woolwine BJ, Shuo C, Schettler P, Drake DF, Haroon E, Miller AH. A randomized controlled trial of the tumor necrosis factor antagonist infliximab for treatment-resistant depression: the role of baseline inflammatory biomarkers. JAMA Psychiatry. 2013 Jan;70(1):31-41. doi: 10.1001/2013.jamapsychiatry.4. PMID 22945416
- [Background] Harrison NA, Brydon L, Walker C, Gray MA, Steptoe A, Critchley HD. Inflammation causes mood changes through alterations in subgenual cingulate activity and mesolimbic connectivity. Biol Psychiatry. 2009 Sep 1;66(5):407-14. doi: 10.1016/j.biopsych.2009.03.015. Epub 2009 May 7. PMID 19423079
- [Background] Hepgul N, Cattaneo A, Agarwal K, Baraldi S, Borsini A, Bufalino C, Forton DM, Mondelli V, Nikkheslat N, Lopizzo N, Riva MA, Russell A, Hotopf M, Pariante CM. Transcriptomics in Interferon-alpha-Treated Patients Identifies Inflammation-, Neuroplasticity- and Oxidative Stress-Related Signatures as Predictors and Correlates of Depression. Neuropsychopharmacology. 2016 Sep;41(10):2502-11. doi: 10.1038/npp.2016.50. Epub 2016 Apr 12. PMID 27067128
- [Background] Carvalho LA, Torre JP, Papadopoulos AS, Poon L, Juruena MF, Markopoulou K, Cleare AJ, Pariante CM. Lack of clinical therapeutic benefit of antidepressants is associated overall activation of the inflammatory system. J Affect Disord. 2013 May 15;148(1):136-40. doi: 10.1016/j.jad.2012.10.036. Epub 2012 Nov 27. PMID 23200297
- [Background] Cattaneo A, Ferrari C, Uher R, Bocchio-Chiavetto L, Riva MA; MRC ImmunoPsychiatry Consortium; Pariante CM. Absolute Measurements of Macrophage Migration Inhibitory Factor and Interleukin-1-beta mRNA Levels Accurately Predict Treatment Response in Depressed Patients. Int J Neuropsychopharmacol. 2016 Sep 30;19(10):pyw045. doi: 10.1093/ijnp/pyw045. Print 2016 Oct. PMID 27207917
- [Background] Vogelzangs N, Beekman AT, van Reedt Dortland AK, Schoevers RA, Giltay EJ, de Jonge P, Penninx BW. Inflammatory and metabolic dysregulation and the 2-year course of depressive disorders in antidepressant users. Neuropsychopharmacology. 2014 Jun;39(7):1624-34. doi: 10.1038/npp.2014.9. Epub 2014 Jan 20. PMID 24442097
- [Background] Benedetti F, Poletti S, Hoogenboezem TA, Locatelli C, de Wit H, Wijkhuijs AJM, Colombo C, Drexhage HA. Higher Baseline Proinflammatory Cytokines Mark Poor Antidepressant Response in Bipolar Disorder. J Clin Psychiatry. 2017 Sep/Oct;78(8):e986-e993. doi: 10.4088/JCP.16m11310. PMID 28922589
- [Background] Dinan TG. Inflammatory markers in depression. Curr Opin Psychiatry. 2009 Jan;22(1):32-6. doi: 10.1097/YCO.0b013e328315a561. PMID 19122532
- [Background] Otte C, Gold SM, Penninx BW, Pariante CM, Etkin A, Fava M, Mohr DC, Schatzberg AF. Major depressive disorder. Nat Rev Dis Primers. 2016 Sep 15;2:16065. doi: 10.1038/nrdp.2016.65. PMID 27629598
- [Background] WHO, 2008 The global burden of disease: 2004 update